CLINICAL TRIAL: NCT01238679
Title: A Phase I, Randomized, Subject and Investigator-Blind, Sponsor Open, Multiple Escalating Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of PF-04958242 in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability and Pharmacokinetics of PF-04958242 in Healthy Adult Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1701002
Record Dates: First submitted 2010-11-02; First posted 2010-11-10 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — PF-04958242

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1 (Experimental): Participants received an oral solution of 0.03 milligrams (mg) of PF-04958242, every 12 hours for 14 days.
  Interventions: Drug: PF-04958242
- Cohort 2 (Experimental): Participants received an oral solution of 0.05 mg of PF-04958242, every 24 hours for 14 days.
  Interventions: Drug: PF-04958242
- Cohort 3 (Experimental): Participants received an oral solution of 0.10 mg of PF-04958242, every 24 hours for 14 days.
  Interventions: Drug: PF-04958242
- Cohort 4 (Experimental): Participants received an oral solution of 0.15 mg of PF-04958242, every 24 hours for 14 days.
  Interventions: Drug: PF-04958242
- Cohort 5 (Experimental): Participants received an oral solution of 0.20 mg of PF-04958242, every 24 hours for 14 days.
  Interventions: Drug: PF-04958242
- Cohort 6 (Experimental): Participants received an oral solution of 0.25 mg of PF-04958242, every 24 hours for 14 days.
  Interventions: Drug: PF-04958242
- Matching Placebo (Placebo Comparator): Participants received an oral solution of matching placebo, every 12 or 24 hours for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04958242 — Administered as specified in the treatment arm
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Matching Placebo

SUMMARY:
The primary objective of this study evaluates the safety and tolerability of multiple, escalating doses of PF-04958242 administered orally to healthy adult participants.This study also evaluates the plasma and urine multiple dose pharmacokinetics (PK) of PF-04958242.

DETAILED DESCRIPTION:
A decision was made to terminate the B1701002 study so that emerging data from the study and from a preclinical study in rats could be further examined and incorporated into a new study design and protocol.

This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kilograms per meter quared (kg/m2);
* Total body weight >50 kilograms (kg) (110 pounds [lbs]);

Key Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing);
* Positive urine drug screen;
* Pregnant or nursing females, and females of child bearing potential;
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11-24 (Actual); Primary Completion 2011-05-03 (Actual); Study Completion 2011-05-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events and Serious Adverse Events | Baseline up to Day 23
  An adverse event is any untoward medical occurrence in a clinical investigation subject administered a product or medical device. A serious adverse event or serious adverse drug reaction is any untoward medical occurrence at any dose that: Results in death; Is life-threatening (immediate risk of death); Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent or significant disability/incapacity; Results in congenital anomaly/birth defect.
Maximum Plasma Drug Concentration (Cmax) for Single Dose | Day 1 and at multiple time points up to Day 17
Time to Reach Maximum Plasma Concentration (Tmax) for Single Dose | Day 1 and at multiple time points up to Day 17
Area Under the Concentration Time-curve During a Dosage Interval (AUCτ) for Single Dose | Day 1 and at multiple time points up to Day 17
Maximum Observed Plasma Concentration (Cmax) for Steady State | Day 1 and at multiple time points up to Day 17
Area Under the Plasma Drug Concentration-Time Curve During a Dosage Interval (AUCτ) for Steady State | Day 1 and at multiple time points up to Day 17
Apparent Total Clearance of the Drug from Plasma (CL/F) for Steady State | Day 1 and at multiple time points up to Day 17
Apparent Volume of Distribution During Terminal Phase (Vz/F) for Steady State | Day 1 and at multiple time points up to Day 17
Elimination Half-Life (t1/2) for Steady State | Day 1 and at multiple time points up to Day 17
Accumulation Ratio (AUC(τ,ss)/AUC(τ,sd)) for Steady State | Day 1 and at multiple time points up to Day 17
Percent of Dose Eliminated in Urine Unchanged (Ae%) | Day 14
Amount of PF-04958242 Eliminated in Urine Unchanged (Ae) | Day 14
Renal Clearance (CLr) | Day 14
Time to Reach Maximum Plasma Concentration (Tmax) for Steady State | Day 1 and at multiple time points up to Day 17

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Singapore, Singapore